CLINICAL TRIAL: NCT00658554
Title: Bioequivalence Study of ARQ 197 Amorphous and Crystalline Polymorphs A and B in Normal Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ArQule, Inc., a subsidiary of Merck Sharp & Dohme LLC, a subsidiary of Merck & Co., Inc. (Rahway, NJ USA) (Industry)
Responsible Party: Nigel Rulewski, MD Chief Medical Officer, ArQule
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: ARQ 197-113
Expanded Access: Available
Record Dates: First submitted 2008-04-11; First posted 2008-04-15 (Estimated); Last update posted 2008-06-19 (Estimated); Status verified 2008-06

CONDITIONS: Healthy
MeSH Terms: interventions — ARQ 197

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ARQ 197 — Treatment with ARQ 197

SUMMARY:
This is a bioequivalence study designed to compare three solid states of ARQ 197 in normal healthy volunteers using a randomized crossover design.

DETAILED DESCRIPTION:
This is a bioequivalence study designed to compare three solid states of ARQ 197 in normal healthy volunteers using a randomized crossover design.

The primary objective is to obtain pharmacokinetic data to assess bioequivalence among three solid states of ARQ 197: amorphous, crystalline polymorph A and crystalline polymorph B.

ELIGIBILITY:
Inclusion Criteria:

* Subject must provide written informed consent prior to any study related procedures
* Subjects must be between the ages of 18 and 65 years
* Male participants must have been surgically sterilized
* Female participants must have been surgically sterilized or be post menopausal and must have a negative serum pregnancy test
* All participants will be phenotypically extensive metabolizers based on their CYP C19 genotype.

Exclusion Criteria:

* Males who are not surgically sterilized
* Females of child-bearing potential who are not surgically sterilized
* Any clinically significant acute or unstable physical or psychological disease based on medical history or screening physical examination
* Any clinically significant abnormality in the screening laboratory tests or ECG
* Received any investigational drugs within four weeks
* Human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV) infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-04; Primary Completion 2008-05 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
To obtain pharmacokinetic data to assess bioequivalence among three solid states of ARQ 197: amorphous, crystalline polymorph A and crystalline polymorph B. | May 2008

SECONDARY OUTCOMES:
To monitor safety of the three solid states of ARQ 197. | May 2008

CONTACTS AND LOCATIONS:
Overall Officials: Ronald M Kimberlin, MD, Principal Investigator — Covance Clinical Research Unit
Locations (1):
- Covance Clinical Research Unit, Inc., Evansville, Indiana, United States